CLINICAL TRIAL: NCT05719961
Title: Bioequivalence Studyof INS062 Injection and NovoRapid ®in Healthy Subjects and Pharmacokinetics and Pharmacodynamics Study of Single Subcutaneous Injection of HR20014 in Healthy Subjects
Brief Title: Bioequivalence Study of INS062 and Pharmacokinetics and Pharmacokinetics Study of Single Injection of HR20014 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR20014-101
Record Dates: First submitted 2023-01-28; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- INS062 (Experimental)
  Interventions: Drug: INS062 injection
- NovoRapid ® (Active Comparator)
  Interventions: Drug: Insulin Aspart
- HR20014 (Experimental)
  Interventions: Drug: HR20014 injection
- BIAsp 30 (Active Comparator)
  Interventions: Drug: Insulin Aspart 30 Injection

INTERVENTIONS:
Drug: INS062 injection — Part I: A single dose of 1.2noml/kg is administered.
  Arms: INS062
Drug: Insulin Aspart — Part I: A single dose of 0.2U/kg is administered.
  Arms: NovoRapid ®
Drug: HR20014 injection — Part II: Ascending single doses at three dose levels
  Arms: HR20014
Drug: Insulin Aspart 30 Injection — Part II: A single dosewas administered
  Arms: BIAsp 30

SUMMARY:
This study was divided into two parts. The aim of this study is to investigate the bioequivalence of INS062 injection andNovoRapid ® in healthy subjects(Part I), and to investigate the pharmacokinetics and pharmacodynamics of single dose of HR20014 injection and BIAsp 30 in healthy subjects(Part II).

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged 18 ~ 45 (including the boundary. value)(Part I). Subjects aged 18 ~ 45 (including the boundary value), male or female(Part II).
2. Subjects who are considered to be generally healthy, based on an assessment of medical history, physical examination and clinical laboratory data, as judged by the Investigator
3. Body Mass Index (BMI) between 18.0-26.0 kg/m2 (both inclusive).

Exclusion Criteria:

1. A history of recurrent or severe drug food allergy, or known or suspected allergy to any component of the study drug.
2. Have a history of hypertension.
3. Severe systemic infectious diseases within 1 month before screening.
4. Use of prescription drugs (topical eye/nasal drops and creams and occasional antipyretic and analgesic drugs such as acetaminophen within recommended doses are permitted) and over-the-counter drugs, and Chinese herbal medicine (regular vitamins are allowed) within 2 weeks before screening.
5. Presence of any abnormal and clinically significant laboratory tests.
6. 12-lead electrocardiogram (ECG) showed abnormal and clinically significant.
7. Known or suspected history of drug abuse or positive urine drug screening test within screening period.
8. Those who have participated in any drug clinical trials within 3 months or 5 half-life periods before screening (The elder shall prevail), who participated in clinical trials are defined as random, prior to screening;
9. Women who are pregnant, breastfeeding or planning to conceive, or women of childbearing potential (WOCBP) are reluctant to use appropriate contraception during the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve （Part I） | 0 to 10 hours after dosing
  Linear Up Log Down
Maximum concentration（Part I） | 0 to 10 hours after dosing
  Observed value
Area under the Glucose Infusion Rate (GIR) - time curve （Part I） | 0 to 10 hours after dosing
  Based on smoothed data
Maximum GIR （Part I） | 0 to 10 hours after dosing
  Based on smoothed data
Area under the Glucose Infusion Rate (GIR) - time curve （Part II） | 0h to 24 hours after dosing
  Based on smoothed data
Maximum GIR（Part II） | 0 to 24 hours after dosing
  Based on smoothed data
Time to maximum GIR （Part II） | 0 to 24 hours after dosing
  Based on smoothed data
Area under the concentration-time curve （Part II） | 0 to 120 hours after dosing
  Linear Up Log Down
Maximum concentration（Part II） | 0 to 120 hours after dosing
  Observed value
Time to maximum concentration （Part II） | 0 to 120 hours after dosing
  Observed value

SECONDARY OUTCOMES:
Time to maximum concentration （Part I） | 0 to 10 hours after dosing
  Observed value
Terminal half-life （Part I） | 0 to 10 hours after dosing
  Terminal half-life of insulin aspart
Time to maximum GIR （Part I） | 0 to 10 hours after dosing
  Based on smoothed data
Incidence of anti-drug antibody (ADA)（Part I） | from 0 hour after dosing to 3-14 days after the last dose
  Incidence of ADA for insulin aspart
Incidence and severity of adverse events (AEs)（Part I） | from screening to 3-14 days after the last dose
  The safety of test drug will be assessed
Incidence of anti-drug antibody (ADA)（Part II） | from 0 hour to 7-21 days after the last dose
Incidence and severity of adverse events (AEs)（Part II） | from screening to 7-21 days after the last dose
  The safety of test drug will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided